CLINICAL TRIAL: NCT07317154
Title: A Phase 1 Study Of The Safety And Immunogenicity Of Peptide-loaded Autologous Dendritic Cell Vaccination In Recurrent Respiratory Papillomatosis (RRP) Patients
Brief Title: Autologous Dendritic Cell Vaccine For Recurrent Respiratory Papillomatosis (RRP) Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David G. Lott, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-002592
Record Dates: First submitted 2025-12-01; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Respiratory Papillomatosis
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Disease Group (Experimental): Patients with clinically confirmed human papilloma virus (HPV)6+ Recurrent Respiratory Papillomatosis (RRP) in the laryngeal mucosa at the time of recruitment and patients with records of RRP in laryngeal mucosa at least once in the past 6-12 months at the time of recruitment.
  Interventions: Biological: Immunotherapy

INTERVENTIONS:
Biological: Immunotherapy — Each patient will receive 5 doses autologous immunotherapy intradermally.
  Other Names: Autologous HPV6 E6-and E7-derived peptide-loaded dendritic cell

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of autologous DC vaccine in recurrent respiratory papillomatosis patients

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of recurrent respiratory papillomatosis.
* Patients with papillomas in the laryngeal mucosa at the time of recruitment and patients with records of recurrent papillomas in laryngeal mucosa at least once in the past 6-12 months at the time of recruitment. NOTE: The presence of papillomas in laryngeal mucosa or clinical records of the presence of papillomas in laryngeal mucosa is required.
* Human papilloma virus (HPV)6+ RRP in larynx
* ECOG (Eastern cooperative oncology group performance test) performance status 0 or 1 (Appendix I).
* The following laboratory values obtained ≤ 28 days prior to apheresis.

  * Absolute neutrophil count (ANC) ≥1.0 x 109 /L
  * Platelet count (PLT) ≥ 75 x 109 /L
  * Hemoglobin ≥ 8.5 g/dL
  * Lymphocytes ≥ 0.3 x 109 /L
  * Total bilirubin ≤ 2 x upper limit of normal (ULN), unless patient has a documented history of Gilbert's disease, then Direct bilirubin ≤1.0 mg/dL.
  * Aspartate transaminase (AST) ≤ 3 x ULN
  * Creatinine ≤ 2.0 mg/dL
  * Monocytes ≥ 0.25 x 109 /L
* Able to provide informed written consent.
* Willingness to return to Mayo Clinic Arizona for follow-up appointments
* Willingness to provide blood samples for immune assessment and other tests
* Willingness to provide papilloma tissues that will be surgically removed
* Agree that during the trial, male participants will not father a child and female participants cannot be or become pregnant if they are of child-bearing potential.
* Subjects must fulfill one of the following conditions:

  * Agree to use one highly effective or combined contraceptive method that results in a failure rate of methods must always be supplemented with the use of spermicide.
  * Be surgically sterile (vasectomy in males or absence of ovaries and/or uterus in females).
  * Be of non-childbearing potential (≥12 months of non-therapy-induced amenorrhea, confirmed by follicle stimulating hormone [FSH], if not on hormone replacement).

Exclusion Criteria:

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other approved or investigational agent (including immune checkpoint blockers, immune modulators, and therapeutic vaccine models) for recurrent respiratory papillomatosis patients which would be considered as a treatment for the papillomas in laryngeal mucosa ≤ 6 months prior to study enrollment.
* Other active malignancy ≤ 5 years prior to enrollment. NOTE: If there is a history or prior malignancy, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin, they must not be receiving other specific treatment for their cancer within one year.
* History of unstable heart disease including myocardial infarction ≤ 6 months prior to registration, congestive heart failure requiring use of ongoing maintenance therapy, significant cardiac dysfunction (left ventricular injection fraction 24 hours) documented by repeated measurement ≤ 4 weeks prior to registration
* Diagnosis of autoimmune disease, including, but not limited to, systemic lupus erythematosus, multiple sclerosis, rheumatoid arthritis, or ankylosing spondylitis.
* Use of a systemic steroid (> 5 mg prednisone daily or equivalent) ≤ 4 weeks prior to registration.
* Pregnant or breastfeeding or planning on becoming pregnant during the study period.
* Requirement for central line placement for cell collections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 20 months
  Safety will be assessed as number of participants to experience adverse events, including systemic symptoms, irritation, inflammation, and any adverse events identified through physical exam and blood counts.

SECONDARY OUTCOMES:
Papilloma Resolution | 20 months
  To evaluate the absence of laryngeal papilloma we will measure the number of laryngeal papilloma at completion of the treatment. This measurement will be compared to 3-year baseline data, or shorter based on date of diagnosis, for each patient as a self-control to interpret time and severity of recurrence.
Time to Disease Recurrence | 20 months
  To measure time to disease recurrence of patients treated with autologous immunotherapy, we will measure the number of laryngeal papilloma during the treatment. This measurement will be compared to 3-year baseline data, or shorter based on date of diagnosis, for each patient as a self-control to interpret time and severity of recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: David G Lott, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials